CLINICAL TRIAL: NCT05728424
Title: ONE WEEK VS. TWO WEEKS VONOPRAZAN CONTAINING TRIPLE REGIMEN FOR ERADICATION OF HELICOBACTER PYLORI:
Brief Title: One vs Two Weeks Treatment for H.Pylori Eradication A RANDOMIZED NON-INFERIORITY PLACEBO CONTROLLED TRIAL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Collaborators: Searle Pharmaceuticals (Unknown)
Responsible Party: Principal Investigator, SHAHAB ABID, Professor Of Medicine, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-7002-21047
Record Dates: First submitted 2023-01-09; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Amoxicillin; Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2 weeks vonoprazan containing triple regimen (Active Comparator): For two weeks:
  Vonaprazan: 20 mg twice daily Amoxicillin: 1gm twice daily Levofloxacin: 500 mg once daily
  Interventions: Drug: Vonoprazan, Amoxicillin, Levofloxacin
- 1 week vonoprazan containing triple regimen (Placebo Comparator): For One week:
  Vonaprazan: 20 mg twice daily Amoxicillin: 1gm twice daily Levofloxacin: 500 mg once daily
  For the second week:
  Placebo
  Interventions: Drug: Vonoprazan, Amoxicillin, Levofloxacin

INTERVENTIONS:
Drug: Vonoprazan, Amoxicillin, Levofloxacin — No additional information

SUMMARY:
1. To assess the efficacy of the duration of Vonoprazan based triple regimen (one versus two weeks), in the eradication of H-pylori among patients attending gastroenterology clinics of Karachi, Pakistan.
2. To assess the improvement in the quality of life of patients receiving Vonoprazan as part of the triple regimen.

DETAILED DESCRIPTION:
Introduction: The overall aim of the study is to assess the efficacy of one week of Vonoprazan compared to two weeks of Vonoprazan in eradicating H-Pylori in patients with dyspeptic symptoms.

H. pylori is a pathogenic Gram-negative spiral bacillus that survives in the acid environment of the stomach. It is a leading cause of chronic gastritis, peptic ulcers, non-ulcer dyspepsia, gastric adenocarcinoma and mucosa-associated lymphoid tissue (MALT) lymphoma. It is estimated that up to 50% of the total world population are infected with H. pylori. The prevalence of H. Pylori infection is currently rising in the developing world. Modified one-week triple therapy (two antibiotics for a week and a potassium-competitive acid blocker for 4-8 weeks) represents the most advanced prescribed regimen for H. pylori infection. With current and widely used therapeutic regimens, (such as two antibiotics and a proton pump inhibitor) there is a significant failure rate for the eradication of microorganism. Therefore, interventions that can improve H-pylori eradication along with improving patient's quality of life are highly important.

Vonoprazan is a potassium-competitive acid blocker, which inhibits the H+/K+ pump in the stomach. Unlike proton pump inhibitors, Vonoprazan inhibits the pump in a competitive and reversible manner. Hence, it is expected to be at least as effective as PPIs in the elimination of Helicobacter Pylori. Assessing the duration of Vonoprazan based triple therapy is of great concern.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* H pylori infection confirmed by any of the 3 tests C-urea breath test (UBT), , rapid urease test, and stool H pylori antigen.

Exclusion Criteria:

* acute gastrointestinal disease (e.g., acute diarrhea)
* chronic gastrointestinal disease (e.g., inflammatory bowel disease, celiac disease)
* known renal and/or liver failure
* no known malignancy
* varices bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of triple therapy in eradication of H.pylori (based on duration) | 6 months
  a) To assess the efficacy of the duration of Vonoprazan based triple regimen (one versus two weeks), in the eradication of H-pylori among patients attending gastroenterology clinics of Karachi, Pakistan.
  The eradication of H.pylori will be tested using the Urea breath test 6 weeks post treatment.

SECONDARY OUTCOMES:
Quality of life assessment using QoLRAD (quality of life in reflux and dyspepsia) | 6 months
  b) To assess the improvement in the quality of life of patients receiving Vonoprazan as part of the triple regimen.

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided